CLINICAL TRIAL: NCT06981195
Title: Neurofunctional Phenotyping to Investigate the Role of the Orexin System at the Intersection of Opioid Use Disorder and Insomnia Among Women and Men Receiving Buprenorphine
Brief Title: Effects of Lemborexant on Insomnia and Its Relationship to Mood and Behavior on Opioid Use Disorder Subjects
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: HM20031777; R01DA059483 (NIH)
Record Dates: First submitted 2025-05-12; First posted 2025-05-20 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Opioid Use Disorder; Opioid Use; Insomnia; Orexin Antagonist
Keywords: buprenorphine; lemborexant
MeSH Terms: conditions — Opioid-Related Disorders; Sleep Initiation and Maintenance Disorders | interventions — lemborexant

STUDY DESIGN:
Intervention Model Description: double-blind randomized clinical trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Subjects who are randomized to placebo will receive identical capsules to the test product, administered orally.
  Interventions: Drug: Placebo
- Lemborexant (Experimental): Lemborexant (trade name Dayvigo), 10mg capsules, administered orally
  Interventions: Drug: Lemborexant 10 MG

INTERVENTIONS:
Drug: Placebo — Subjects who are randomized to placebo will receive identical capsules to the study drug. During the 8-week intervention phase, participants will be instructed to take one capsule daily, approximately 5-30 minutes before going to bed
  Arms: Placebo
Drug: Lemborexant 10 MG — During the 8-week intervention phase, participants will be instructed to take one capsule daily, approximately 5-30 minutes before going to bed
  Arms: Lemborexant

SUMMARY:
The goal of this clinical trial is to learn about how certain medications used to treat insomnia (e.g., Lemborexant) impact sleep, mood, and behavior in men and women with Opioid Use Disorder who are taking prescribed buprenorphine. The main questions it aims to answer are:

1. What is the effect of the study drug (lemborexant) on sleep outcomes?
2. What is the effect of the study drug (lemborexant) on impulsive behavior (as measured by computer test performance)?
3. What is the effect of the study drug (lemborexant) on mood and other behavior?

Researchers will compare lemborexant to placebo (e.g., sugar pill) to see if participants assigned to 8 weeks of treatment with lemborexant have greater improvements on the measures listed above.

Participants will take the study medication (or placebo) each night for 8 weeks and be asked to come for a total of 23 study visits. Most of these visits will be very short (15-30 minutes). The longer visits will include the screening visit (about 2-3 hrs), baseline visit (about 2.5 hrs), and the post-medication visit (about 2 hrs). Study visits will include things like taking surveys about sleep, drug use, and mood, completing urine drug testing, checking vital signs (e.g., blood pressure), and completing interviews with the study staff. Participants will also be asked to provide two blood samples (one during screening and one after taking the medication). For three two-week periods, participants will be asked to wear a watch to track sleep at home, and to keep a log of sleep and wake times.

ELIGIBILITY:
Inclusion Criteria:

1. Be 18 + years-of-age
2. Meet current DSM-5 criteria for opioid use disorder (OUD) with at least moderate severity
3. Receiving outpatient treatment for OUD with sublingual buprenorphine film/tablets ranging 8mg to 24mg or with extended-release injectable buprenorphine
4. Stabilized on current buprenorphine dosage for at least 4 weeks without intention for dose change within next 3 months.
5. Screening urine toxicology positive for buprenorphine and an appropriate norbuprenorphine level as determined by a study clinician
6. A screening urine toxicology negative for non-prescribed substances (except cannabinoids) with a negative breath (or oral fluid) alcohol screen
7. Screen positive for chronic insomnia on the Insomnia Symptom Questionnaire (ISQ)
8. Have an Insomnia Severity Index score at screening and baseline of 13 or higher
9. Have no clinically significant medical or psychiatric disorder or condition, based on physical exam and medical history performed by study clinician, that in the judgement of the investigator would prevent participation or heighten safety risks
10. Understand the study procedures and provide written informed consent in English language
11. Access to necessary resources for completing virtual surveys and monitoring (i.e., computer or smartphone, internet or cell service)

Exclusion Criteria:

1. Current diagnosis of sleep-related breathing disorder, narcolepsy, somnambulism, or sleep paralysis
2. A positive screen for sleep apnea by the following: Sleep Disorders Screening Battery (STOP-BAG >5) OR home sleep apnea test using WatchPAT with Apnea Hypopnea Index (AHI) with 3% drop in oxygen saturation > 10 OR >50% of respiratory events being central if AHI is between 5-10 OR Oxygen Desaturation < 88% for > 10 minutes, OR oxygen desaturation index (ODI) using 3% drop in oxygen saturation > 10
3. Currently receiving treatment for insomnia (behavioral or pharmacologic)
4. Currently taking a medication to treat a sleep-related condition (e.g., zolpidem) or unable to discontinue over-the-counter drug or supplement used to treat sleep-related condition
5. Currently taking benzodiazepines or other CNS active medications that may increase risk to the participant, per PI discretion (e.g., opioids other than buprenorphine, antipsychotics)
6. Current DSM-5 diagnosis (any severity) of alcohol or drug use disorder (e.g., benzodiazepine, stimulant) with non-prescribed substance use within last 3 months; nicotine use disorder is not considered exclusionary
7. Cannabis use > 3 days/week
8. Uncontrolled serious psychiatric disorder that would make study participation unsafe (such as Bipolar I Disorder, ADHD, Schizophrenia, schizoaffective disorders, major depressive disorder with psychotic features, or a neurological disorder).
9. Uncontrolled neurological, cardiovascular, or pulmonary medical condition such as seizure disorder, recent myocardial infarction, stroke, hospitalization for chronic obstructive pulmonary disease
10. Baseline ECG with clinically significant abnormal conduction or with QTc of greater than 450ms
11. Significant current suicidal or homicidal ideation (C-SSRS "yes" answers on questions 4 or 5) or a history of suicide attempt within the past 6 months
12. Any of the following lab abnormalities: ALT/AST 2 or more times the upper limit of normal, Total bilirubin 2 or more times the upper limit of normal, Creatinine 1.5 or more times the upper limit of normal
13. Pregnant or breastfeeding; Females who are having sex that includes penile penetration must be non-pregnant, non-lactating, and either be of non-childbearing potential (e.g., sterilized via hysterectomy, bilateral tubal ligation, or bilateral oophorectomy, or at least 1 year post-menopausal) or of childbearing potential, and agree to use an acceptable form of contraception (e.g., IUD, hormonal implant, hormonal patch/ring/pill, condoms (male or female), etc.)
14. Currently taking prescription or over-the counter drugs or dietary supplements known to significantly inhibit CYP3A4 (such as clarithromycin, telithromycin, nefazodone, itraconazole, ketoconazole, atazanavir, darunavir, indinavir, lopinavir, nelfinavir, ritonavir, saquinavir, tipranavir); or CYP3A4 inducers (such as phenobarbital, phenytoin, rifampicin, St. John's Wort, and glucocorticoids)
15. Currently taking lemborexant or any previous medically adverse reaction to lemborexant or other dual orexin receptor antagonists
16. Currently incarcerated or pending incarceration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-27 (Actual); Primary Completion 2029-07-30 (Estimated); Study Completion 2029-07-30 (Estimated)

PRIMARY OUTCOMES:
Insomnia | from baseline to end of 8-week treatment
  Insomnia Severity Index will be used for assessing insomnia related symptoms. Scores on this measure range from 0-28, with higher scores indicating greater symptoms. Mean ISI score per group at baseline and at the end of 8-week treatment will be reported.
Impulsivity | from baseline to end of 8-week treatment
  Impulsive responding will be measured by performance on the 5-trial adjusting delay discounting task, with the outcome being a derived discounting rate. Mean delay discounting rate per group at baseline and at the end of 8-week treatment will be reported.

SECONDARY OUTCOMES:
Insomnia related daily sleep metrics: Total sleep time (TST) | from baseline to end of 8-week treatment
  Total sleep time (TST) will be derived from actigraphy measured by an actigraphy watch. The descriptive statistics of derived TST score per group at baseline and end of 8-week treatment will be reported.
Insomnia related daily sleep metrics: Wake After Sleep Onset (WASO) | from baseline to end of 8-week treatment
  Wake After Sleep Onset (WASO), will be derived from actigraphy measured by an actigraphy watch. The descriptive statistics of derived WASO score per group at baseline and end of 8-week treatment will be reported.
Insomnia related daily sleep metrics: Sleep efficiency (SE) | from baseline to end of 8-week treatment
  Sleep efficiency (SE) will be derived from actigraphy measured by an actigraphy watch. The descriptive statistics of derived SE score per group at baseline and end of 8-week treatment will be reported.
Insomnia related daily sleep metrics: Sleep onset latency (SOL) | from baseline to end of 8-week treatment
  Sleep onset latency (SOL) will be derived from actigraphy measured by an actigraphy watch. The descriptive statistics of derived SOL score per group at baseline and end of 8-week treatment will be reported.
Negative Emotionality: Distress Tolerance Scale (DTS) | from baseline to end of 8-week treatment
  The Distress Tolerance Scale will be used as a measure of negative emotionality. The DTS is a 15-item, 5-point Likert scale measure with item scores ranging from 1-5. Lower scores indicate greater distress tolerance. Mean DTS score per group at baseline and at the end of 8-week treatment will be reported.
Negative Emotionality: Patient Health Questionnaire (PHQ-9) | from baseline to end of 8-week treatment
  The PHQ-9 is a brief (9-item) measure of depressive symptoms. Scores range from 1-27, with higher scores indicating greater severity of depressive symptoms. Mean PHQ-9 score per group at baseline and at the end of 8-week treatment will be reported.
Negative Emotionality: General Anxiety Disorder (GAD-7) | from baseline to end of 8-week treatment
  The GAD-7 is a brief (7-item) measure of anxiety symptoms. Scores range from 0-21, with higher scores indicating greater severity of anxiety symptoms. Mean GAD-7 score per group at baseline and at the end of 8-week treatment will be reported.
Metacognition: Metacognitions Questionnaire (MCQ-30) | from baseline to end of 8-week treatment
  The MCQ-30 a brief (30-item) measure of metacognition. Total scores range from 30-120, with higher scores indicating greater magnitude of problematic metacognitions. Mean MCQ-30 score per group at baseline and at the end of 8-week treatment will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Caitlin E Martin, MD, Principal Investigator — Virginia Commonwealth University Institute for Drug and Alcohol Studies
Locations (1):
- VCU Institute for Drug and Alcohol Studies, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Marcus MM, Alattar M, Chen S, Sabo R, Pignatello T, Ruddley J, Green AR, Swan K, Keyser-Marcus L, Moeller FG, Martin CE. Neurofunctional phenotyping to investigate the role of the orexin system at the intersection of opioid use disorder and insomnia: a protocol for a randomised, placebo-controlled clinical trial of lemborexant in patients with insomnia receiving buprenorphine. BMJ Open. 2025 Oct 28;15(10):e108613. doi: 10.1136/bmjopen-2025-108613. PMID 41151943

DOCUMENTS (1):
  • Informed Consent Form (2025-04-09): https://cdn.clinicaltrials.gov/large-docs/95/NCT06981195/ICF_000.pdf